CLINICAL TRIAL: NCT06021587
Title: Interest of Levosimendan Preconditioning for Cardiac Surgery Under CEC in Heart Failure Patients With Impaired Ejection Fraction
Acronym: LevoCV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Klein Thomas, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023_PI_084
Record Dates: First submitted 2023-07-26; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Levosimendan; Cardiac Surgery; Heart Failure With Reduced Ejection Fraction
Keywords: Levosimendan; Cardiac Surgery; Cardiopulmonary Bypass; Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — Simendan; Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Levosimendan: Major patients in heart failure with impaired LVEF (< 40%) who have undergone left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation between 01/01/2018 and 28/02/2022 at different French Hospital, and who have received Levosimendan preoperatively
  Interventions: Drug: Levosimendan
- Control - No Levosimendan: Major patients in heart failure with impaired LVEF (< 40%) who have undergone left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation between 01/01/2018 and 28/02/2022 at different French Hospital and who have not received Levosimendan preoperatively
  Interventions: Drug: No Levosimendan

INTERVENTIONS:
Drug: Levosimendan — Initiation of levosimendan 48 hours before surgery
  Other Names: Interventional
  Groups: Levosimendan
Drug: No Levosimendan — Without Levosimendan Infusion
  Other Names: Control
  Groups: Control - No Levosimendan

SUMMARY:
Levosimendan, a drug with inotropic, vasodilatory and myocardial protective properties, has been proposed for the prevention and treatment of postoperative low cardiac output syndrome in cardiac surgery. Despite preliminary studies with promising results, large randomized controlled trials aimed at demonstrating the benefits of levosimendan did not show superiority over placebo in this indication. However, in these studies, the infusion was neither performed at the maximum dosage nor during the 24 hours preceding the surgery, but mainly at the very beginning of the operation. However, post hoc analyses showed a reduction in mortality and in the occurrence of low cardiac output syndrome in the subgroup of patients who had undergone isolated coronary artery bypass grafting, in contrast to those who had undergone valvular or combined surgery. Another recent study suggests that under similar conditions, preconditioning with levosimendan started 48 hours before surgery reduces the length of stay in intensive care and the average cost of hospitalization. There are no formal recommendations on the prophylactic use of levosimendan in cardiac surgery for heart failure patients with impaired LVAS. However, the France-Levo registry, a multicenter observational study requested by the HAS, has shown that in real practice there is a place for preconditioning with levosimendan, which is used in this indication for 7% of the patients in the registry. The Cardiovascular Surgery and Transplantation Department of the Nancy Brabois University Hospital, which actively participated in the France-Levo registry, is one of the cardiac surgery centers that uses this practice, as is the University Hospital of Rouen. It is interesting to be able to evaluate retrospectively whether levosimendan preconditioning has a positive impact on the postoperative prognosis of patients and more particularly on the reduction of the length of stay in critical care and in hospital compared to standard management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart failure impaired LVEF (< 40%), who have undergone left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation between 01/01/2018 and 28/02/2022 at different University Hospital in France

Exclusion Criteria:

* Initiation of levosimendan > 48 hours or < 24 hours before surgery ECMO pre- or post-op

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Preoperative heart failure patients with impaired LVEF who underwent left heart surgery (coronary artery bypass grafting and/or mitral and/or aortic valve replacement) under extracorporeal circulation from 01/09/2018 to 28/02/2022 at different University Hospital in France
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) criteria at 30 days | 30 days after Levosimendan exposure
  to evaluate the impact of preconditioning with Levosimendan prior to scheduled cardiac surgery with extracorporeal circulation in patients with heart failure and impaired LVEF on the rate of cardiovascular events at 30 days post-op.

SECONDARY OUTCOMES:
major renal events (MAKE) at 30 days from the date of surgery | 30 days after Levosimendan exposure
  to evaluate the impact of preconditioning with Levosimendan prior to scheduled cardiac surgery under extracorporeal circulation in patients with heart failure and impaired LVEF on the rate of renal events at 30 days post cardiac surgery.
On 1-year mortality | 1 year after Levosimendan exposure
  To evaluate the impact of preconditioning with Levosimendan before cardiac surgery in patients with heart failure and impaired left ventricular dysfunction on 1-year mortality
Length of stay in ICU | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of levosimendan preconditioning preoperatively for cardiac surgery on critical care length of stay in patients with heart failure with impaired preoperative LVAS
the total length of hospital stay | start date of hospitalization in intensive care to the date of discharge from conventional sectors evaluated up to 3 months
  To evaluate the impact of preconditioning with Levosimendan preoperatively for cardiac surgery in patients with heart failure with impaired preoperative left ventricular dysfunction on the total length of hospital stay
Measurement of left ventricular ejection fraction by cardiac ultrasound at hospital discharge | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of Levosimendan preconditioning before cardiac surgery in patients with heart failure and impaired on left ventricular systolic function (measured by cardiac ultrasound) at hospital discharge
duration of catecholamine use after surgery | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of preconditioning with Levosimendan before cardiac surgery in patients with heart failure and impaired left ventricular function before surgery on the duration of catecholamine use after surgery
severity of postcardiotomy cardiogenic shock and/or postoperative vasoplegia using the score Vasoactive Inotropic Score (VIS) | date of start of intensive care hospitalization to date of discharge from intensive care hospitalization assessed up to 3 months
  To evaluate the impact of preconditioning with Levosimendan in preoperative cardiac surgery in patients with heart failure with impaired preoperative LVAS on the severity of postcardiotomy cardiogenic shock and/or postoperative vasoplegia. High VIS was empirically defined as ≥ 20. Maximum VIS≥20 predicts an increased likelihood of a poor composite clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Thomas KLEIN, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- 'CHRU Nancy, Vandœuvre-lès-Nancy, Meurthe Et Moselle, France

IPD SHARING:
Plan to Share IPD: Undecided